CLINICAL TRIAL: NCT01472588
Title: Translating the DPP Lifestyle Intervention to Rural African-American Communities
Brief Title: Translating the Diabetes Prevention Program (DPP) Lifestyle Intervention to Rural African-American Communities (HEALTHY Ways)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UAMS IRB#: 99099; 5P20MD002329 (NIH)
Record Dates: First submitted 2011-10-25; First posted 2011-11-16 (Estimated); Last update posted 2023-10-23 (Actual); Status verified 2014-09

CONDITIONS: Overweight
MeSH Terms: conditions — Overweight | interventions — CD5L protein, human; United States Dept. of Health and Human Services

ARMS (3):
- Community Health Coach (Experimental): DPP behavioral lifestyle intervention delivered by Community Health Coach (CHWs)
  Interventions: Behavioral: DPP lifestyle intervention-Community Health Coach (CHWs)
- Public Health Coach (Experimental): DPP behavioral lifestyle intervention delivered by health professionals (PHCs)
  Interventions: Behavioral: DPP Lifestyle intervention--health professionals/(PHCs)
- Self Help (Other): Booklet, Aim for a Healthy Weight (DHHS, NIH-NHLBI) provided.
  Interventions: Other: Self Help

INTERVENTIONS:
Behavioral: DPP lifestyle intervention-Community Health Coach (CHWs) — Lifestyle counseling. During a 16 month period, the behavioral weight loss program (n=24 sessions of the DPP lifestyle intervention) is delivered by CHWs in group format in community settings.
  Other Names: DPP Lifestyle Balance Program
  Arms: Community Health Coach
Behavioral: DPP Lifestyle intervention--health professionals/(PHCs) — Lifestyle counseling. During a 16 month period, the behavioral weight loss program (n=24 sessions of the DPP lifestyle intervention) is delivered by PHCs in group format in community settings.
  Other Names: DPP Lifestyle Balance Program
  Arms: Public Health Coach
Other: Self Help — Public education/information booklet on weight management.
  Other Names: Aim for a Healthy Weight (DHHS, NIH-NHLBI); --publically available education material.
  Arms: Self Help

SUMMARY:
Obesity is a significant and growing problem in the US that negatively impacts health and well-being of racial and ethnic minorities, people of low socioeconomic status, and persons living in rural communities and in the South. Obesity is a major concern in Arkansas, where the obesity rate for adults is higher than the rate for other adults in the nation. However effective weight loss programs are not typically available in these communities. Research has shown that the Diabetes Prevention Program (DPP) lifestyle intervention is effective in promoting weight loss in high risk individuals through changes in diet and physical activity that significantly reduce the chances of type 2 diabetes. Effective methods are desperately needed to translate the DPP to community settings, where obesity is a compelling public health burden. A major step in translating the DPP is to examine the efficacy of health professionals and community health workers (CHWs) in delivering the program in real-world settings. This is an important issue from the perspective of how evidence-based weight loss interventions can be provided to underserved, and resource constrained communities that typically may not have access to trained professionals for program delivery. The current project is a 5 year randomized controlled trial that examines DPP delivery and weight outcomes for individuals randomly assigned to either: (1) the DPP intervention delivered by CHWs or (2) the DPP intervention delivered by health professionals or (3) the Self Help condition. The study population consists of overweight adults (body mass index (BMI) > 25) who reside in communities with a high proportion of African Americans. Primary outcome is change in body weight at 16 months. Cost effectiveness and lifestyle behaviors are also evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Non-institutionalized men and women aged 18 and older
2. BMI [weight (kg)/ height (m2)] > 25
3. Able to walk for exercise
4. Able to provide informed consent
5. Willing to accept random assignment

Exclusion Criteria:

1. Currently pregnant or nursing, or pregnant within previous 6 months
2. Recent heart attack or stroke (in past 6 months)
3. Congestive heart failure (NYHA Class 3-4)
4. History of bariatric surgery or weight loss in excess of 10% in past 6 months
5. Current use of weight loss medications
6. Another member of household enrolled in study
7. Presence of significant impairment that might interfere with participation, such as underlying disease likely to limit lifespan, infectious disease (e.g., HIV, tuberculosis), substantial cognitive impairment, renal dialysis, diagnosis of schizophrenia, psychosis or substance abuse, or other condition that might compromise participation or for which weight loss is not recommended
8. Plans to move from the area within the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 277 (Actual)
Dates: Start 2007-09; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Weight Loss | 16 months
  change in weight (% loss) from baseline to 16 months

SECONDARY OUTCOMES:
Physical Activity | 16 months
  change in number of minutes of physical activity, baseline to 16 months.

CONTACTS AND LOCATIONS:
Overall Officials: Theresa E. Prewitt, DrPH, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States